CLINICAL TRIAL: NCT06019910
Title: The Effects of Snus on Home Blood Pressure and Metabolism
Brief Title: Snus and Home Blood Pressure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Fredrik H Nystrom, Professor of internal medicine and endocrinology, University Hospital, Linkoeping
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: snus2023
Record Dates: First submitted 2023-07-30; First posted 2023-08-31 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Blood Pressure; Dyslipidemias; Dysglycemia; Obesity
MeSH Terms: conditions — Dyslipidemias; Obesity | interventions — Tobacco, Smokeless; Tobacco Products

STUDY DESIGN:
Intervention Model Description: At baseline, all participants use snus, and will be asked to quit their usage. They will then be followed for up to 12 weeks. If and when they relapse in snus use, another 12 weeks will commence, during which the same measurements will repeated but for a second period of up to 12 weeks.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Snus with or without tobacco (Experimental): Snus cessation followed by potential snus relapse
  Interventions: Other: Snus with or without tobacco

INTERVENTIONS:
Other: Snus with or without tobacco — At baseline, participants have used the intervention daily for at least 30 days. They will then cease usage of the intervention abruptly. After 3 weeks, they may continue to abstain from the intervention or relapse at their own discretion.

SUMMARY:
Snus is a type of snuff that is administered sublabially, that has not been studied regarding the effects on home blood pressure and metabolism on a longer time frame. The primary aim of this study is to evaluate the effect of snus on home BP within weeks to months in former snus users who continue to not use snus or relapse in daily snus use, respectively. The secondary aim is to evaluate the effects on metabolic measurements. The hypothesis is that BP will increase amongst the participants that resume snus intake.

28 healthy volunteers with a pre-existing daily use of snus will be recruited and followed during snus cessation. Home blood pressure, lipid and metabolic markers will be measured before and after snus cessation, as well as after snus relapse if such a relapse occurs.

DETAILED DESCRIPTION:
Both elevated blood pressure (BP) and cigarette smoking increases the risk of cardiovascular disease. Nicotine, through effects on the nervous system and catecholamine release, increases BP and heart rate, peaking 5-10 minutes after exposure, after which tolerance to nicotine reduces its hemodynamic effects. Smoking also increases energy expenditure, but studies on smoking and long-term metabolism have shown conflicting results.

Snus is a type of snuff that is administered sublabially, that has not been studied regarding the effects on home blood pressure and metabolism on a longer time frame. The primary aim of this study is to evaluate the effect of snus on home BP within weeks to months in former snus users who continue to not use snus or relapse in daily snus use, respectively. The secondary aim is to evaluate the effects on metabolic measurements. The hypothesis is that BP will increase amongst the participants that resume snus intake.

28 healthy volunteers with a pre-existing daily use of snus will be recruited and followed during snus cessation for 3 months. Home blood pressure, lipid and metabolic markers will be measured before and after snus cessation. Furthermore, for participants which relapse in snus use, the same measurements will be followed for an additional 3 months. Home blood pressure will be measured daily, and participants will also report the amount of snus use each day. At week 0, 4 and 12 of snus cessation and snus relapse, the following measurements will also be made: body weight as well as plasma glucose, blood glycated hemoglobin (HbA1c), serum insulin, plasma lipid profile (total cholesterol, low-density lipoprotein, high-density lipoprotein, and triglycerides), plasma hsCRP, plasma creatinine, plasma sodium, and plasma potassium.

As reimbursement, participants will receive (at least) 1000 Swedish krona (Approx 94 US dollar) for the drawing of blood tests. All participants will give written, informed consent prior to participation. The study will comply with the declaration of Helsinki and be approved by the Swedish Ethical Review Authority. Prior to commencement, the study will be registered at ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* daily use (defined as at least once daily for at least 1 month) o snus
* the ability to use online questionnaires written and answered in Swedish

Exclusion Criteria:

* simultaneous use of any other nicotine or tobacco product (including cigarette smoking, e-cigarettes, and nicotine replacement therapy)
* drug use (including cannabis)
* alcohol dependence
* known cardiovascular disease (including hypertension, previous myocardial infarction, stroke, peripheral arterial disease, or angina pectoris), kidney disease, hormonal disease (including diabetes mellitus) or eating disorder
* current or planned pregnancy.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Home blood pressure during snus cessation | 4-12 weeks
  Change in home blood pressure from baseline until week 4 and week 12 respectively
Home blood pressure during snus relapse | 4-12 weeks
  Change in home blood pressure from week 0 of snus relapse until week 4 and week 12 respectively

SECONDARY OUTCOMES:
Body weight during snus cessation | 4-12 weeks
  Change in body weight from baseline until week 4 and week 12 respectively
Concentration of plasma lipids during snus cessation | 4-12 weeks
  Change in plasma lipids from baseline until week 4 and week 12 respectively
Concentration of fasting plasma glucose during snus cessation | 4-12 weeks
  Change in fasting plasma glucose from baseline until week 4 and week 12 respectively
Concentration of fasting plasma insulin during snus cessation | 4-12 weeks
  Change in fasting plasma insulin from baseline until week 4 and week 12 respectively
Concentration of blood HbA1c during snus cessation | 4-12 weeks
  Change in blood HbA1c from baseline until week 4 and week 12 respectively
Body weight during snus relapse | 4-12 weeks
  Change in body weight from week 0 of snus relapse until week 4 and week 12 respectively
Concentration of plasma lipids during snus relapse | 4-12 weeks
  Change in plasma lipids from week 0 of snus relapse until week 4 and week 12 respectively
Concentration of fasting plasma glucose during snus relapse | 4-12 weeks
  Change in fasting plasma glucose from week 0 of snus relapse until week 4 and week 12 respectively
Concentration of fasting plasma insulin during snus relapse | 4-12 weeks
  Change in fasting plasma insulin from week 0 of snus relapse until week 4 and week 12 respectively
Concentration of blood HbA1c during snus relapse | 4-12 weeks
  Change in blood HbA1c from week 0 of snus relapse until week 4 and week 12 respectively

CONTACTS AND LOCATIONS:
Overall Officials: Fredrik H Nyström, PhD, MD, Principal Investigator — Linkoeping University
Locations (1):
- Primary Health Care Center Cityhälsan Centrum, Norrköping, Sweden

REFERENCES:
- [Background] Williams B, Mancia G, Spiering W, Agabiti Rosei E, Azizi M, Burnier M, Clement DL, Coca A, de Simone G, Dominiczak A, Kahan T, Mahfoud F, Redon J, Ruilope L, Zanchetti A, Kerins M, Kjeldsen SE, Kreutz R, Laurent S, Lip GYH, McManus R, Narkiewicz K, Ruschitzka F, Schmieder RE, Shlyakhto E, Tsioufis C, Aboyans V, Desormais I; Authors/Task Force Members:. 2018 ESC/ESH Guidelines for the management of arterial hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension: The Task Force for the management of arterial hypertension of the European Society of Cardiology and the European Society of Hypertension. J Hypertens. 2018 Oct;36(10):1953-2041. doi: 10.1097/HJH.0000000000001940. PMID 30234752
- [Background] Benowitz NL, Pipe A, West R, Hays JT, Tonstad S, McRae T, Lawrence D, St Aubin L, Anthenelli RM. Cardiovascular Safety of Varenicline, Bupropion, and Nicotine Patch in Smokers: A Randomized Clinical Trial. JAMA Intern Med. 2018 May 1;178(5):622-631. doi: 10.1001/jamainternmed.2018.0397. PMID 29630702
- [Background] Middlekauff HR, Park J, Moheimani RS. Adverse effects of cigarette and noncigarette smoke exposure on the autonomic nervous system: mechanisms and implications for cardiovascular risk. J Am Coll Cardiol. 2014 Oct 21;64(16):1740-50. doi: 10.1016/j.jacc.2014.06.1201. PMID 25323263
- [Background] Martinez-Morata I, Sanchez TR, Shimbo D, Navas-Acien A. Electronic Cigarette Use and Blood Pressure Endpoints: a Systematic Review. Curr Hypertens Rep. 2020 Nov 23;23(1):2. doi: 10.1007/s11906-020-01119-0. PMID 33230755
- [Background] Audrain-McGovern J, Benowitz NL. Cigarette smoking, nicotine, and body weight. Clin Pharmacol Ther. 2011 Jul;90(1):164-8. doi: 10.1038/clpt.2011.105. Epub 2011 Jun 1. No abstract available. PMID 21633341
- [Background] Chiolero A, Faeh D, Paccaud F, Cornuz J. Consequences of smoking for body weight, body fat distribution, and insulin resistance. Am J Clin Nutr. 2008 Apr;87(4):801-9. doi: 10.1093/ajcn/87.4.801. PMID 18400700
- [Background] Hofstetter A, Schutz Y, Jequier E, Wahren J. Increased 24-hour energy expenditure in cigarette smokers. N Engl J Med. 1986 Jan 9;314(2):79-82. doi: 10.1056/NEJM198601093140204. PMID 3941694
- [Derived] Af Geijerstam P, Joelsson A, Radholm K, Nystrom FH. Cardiovascular and metabolic changes following 12 weeks of tobacco and nicotine pouch cessation: a Swedish cohort study. Harm Reduct J. 2025 Apr 16;22(1):54. doi: 10.1186/s12954-025-01195-y. PMID 40241094